CLINICAL TRIAL: NCT04135170
Title: Antibiotic Loaded Bone Cement in Prevention of Periprosthetic Joint Infections in Primary Total Knee Arthroplasty: A Register-based Multicenter Randomized Controlled Non-inferiority Trial (Acronym: ALBA Trial)
Brief Title: Antibiotic Loaded Bone Cement in Prevention of Periprosthetic Joint Infections in Primary Total Knee Arthroplasty
Acronym: ALBA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Norwegian Arthroplasty Register (Other Government)
Collaborators: Helse Vest (Other)
Responsible Party: Principal Investigator, Asst. professor Tesfaye Hordofa Leta (Nurse, Postdoc fellow), Associate professor/ postdoc fellowship, The Norwegian Arthroplasty Register
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NorwegianArthroplastyRegister
Record Dates: First submitted 2019-09-20; First posted 2019-10-22 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Register based randomized control trial; Non-inferiority; Total knee arthroplasty; Antibiotic loaded bone cement; Plain bone cement; Antibiotic resistance bacteria; Periprosthetic joint infection; Patient reported outcome measure; Health related quality of life; Pain; Function; Satisfaction; Revision surgery; Primary surgery
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Patients undergoing full-cemented primary TKA in any Norwegian hospitals are eligible for participation irrespectively of the diagnosis leading to TKA. and randomly assigned to receive ALBC (control group) or plain bone cement (experimental group).
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double blinded, non-inferiority register-based multicenter randomized controlled trial study. To ensure blinding of the patients, all patients are operated by the same surgical method and the type of cement is unknown to the patients. In this study, blinding of the surgeon is not possible because the surgeon recognizes the cement type and has to document the type of cement in the registration form. We believe the primary endpoint of this trial is not likely to be influenced by the surgeon knowledge of the cement used in the index surgery. The data analyst will be blinded for groups until the entire trial analysis has been completed to minimize the risk of bias that may be introduced during the statistical analysis because of the selective use and reporting of statistical tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain bone cement (Experimental)
  Interventions: Combination Product: ALBC vs plain bone cement
- Antibiotic loaded bone cement (Active Comparator)
  Interventions: Combination Product: ALBC vs plain bone cement

INTERVENTIONS:
Combination Product: ALBC vs plain bone cement — The patients undergoing full-cemented primary total knee arthroplasty are allocated to either ALBC or plain bone cement and compare the effectiveness of ALBC use vs pain bone cement bone cement without antibiotic) with respect to revision due to PJI one year after primary TKA surgery.

SUMMARY:
Introduction: The current evidence on the efficacy of Antibiotic Loaded Bone Cement (ALBC) in reducing the risk of periprosthetic joint infections (PJI) after primary joint reconstruction is insufficient. In several European countries, the use of ALBC is routine practice unlike in the US where ALBC use is not approved in low-risk patients. It has been claimed that the antibiotic in ALBC increase the risk of aseptic loosening, risk of systemic toxicity, allergic reaction, and bacterial resistance. Therefore we designed a double-blinded (patients and data analysts) pragmatic multicenter register-based randomized controlled non-inferiority trial to investigate the effects of ALBC compared to plain bone cement in primary total knee arthroplasty (TKA).

Methods and analysis: A minimum of 9,172 patients undergoing full-cemented primary TKA will be recruited and equally randomized into the ALBC group and the plain bone cement group. This trial will be conducted in Norwegian hospitals that routinely perform cemented primary TKA. . The primary outcome will be risk of revision surgery due to PJI at 1-year of follow-up. Secondary outcomes will be:

* risk of revision due to any reason including aseptic loosening at 1-, 6-, 10-, and 20-years of follow-up;
* patient related outcome measures (PROMs) like function, pain, satisfaction, and health-related quality of life at 1-, 6-, and 10-years of follow-up;
* risk of changes in the microbial pattern and resistance profiles of organisms cultured in subsequent revisions at 1-, 6-, 10-, and 20-years of follow-up; and
* cost-effectiveness of routine ALBC vs plain bone cement use in primary TKA. We will use 1:1 randomization with random permuted blocks and stratify by participating hospitals to randomize patients to receive ALBC or plain bone cement. Inclusion, randomization, and follow-up will be through the Norwegian Arthroplasty Register.

Ethics and dissemination: The trial has been approved by the Western Norway Regional Committees on Medical and Health Research Ethics (REK-Vest) (reference number: 2019/751/REK vest) dated: 21.06.2019. The trial results will be reported following the Consolidated Standards of Reporting Trials Extension (CONSORT Extension) reporting guideline 2010 statement for non-inferiority trials. The trial results will be reported to the public through national and international scientific conferences, participating hospitals, patient organizations, and peer-reviewed journals.

Discussion: If we find that plain bone cement is non-inferior to the ALBC, it will challenge the routine use of ALBC in primary arthroplasty, due to ecological concerns and costs. However, if routine use of ALBC is associated with a reduced risk of PJI and with minor impact on bacterial resistance, PROMs, and costs, the well-established use of prophylactic ALBC in primary arthroplasty will be supported

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing full-cemented primary TKA irrespective of the diagnosis leading to TKA

Exclusion Criteria:

* any history of infection in the knee, a need for fully stabilized or hinged TKA, a history of allergy to the antibiotics used in the cement, inability or not willing to consent for inclusion in NAR or the trial, and participation in other studies that might have pharmacological interaction with this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9172 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
risk of revision due to PJI | 1-year follow-up

SECONDARY OUTCOMES:
risk of revision due to any reason including aseptic loosening | 1-, 6-, 10-, and 20-years follow-up
risk of changes in the microbial pattern and resistance profiles of organisms cultured in subsequent revisions | 1-, 6-, 10-, and 20-years follow-up
Change in mean scores from baseline function (in activity of daily life) on the Knee injury and Osteoarthritis Outcome Score (KOOS). | 1-, 6-, and 10-years follow-up
Change in mean scores from baselinein in Visual Analog Sale (the scores range from 0 to 100, with 0 indicating the worst possible state and 100 indicating the best possible state) for pain. | 1-, 6-, and 10-years follow-up
Change in mean scores from baseline in EQ-5D-5L for health related quality of life(HRQoL). | 1-, 6-, and 10-years follow-up
Mean scores in Visual Analog Sale ( the scores range from 0 to 100, with 0 indicating the worst possible state and 100 indicating the best possible state) for patient satisfaction. | 1-, 6-, and 10-years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ove Furnes, MD/PhD, Study Chair — The Norwegian Arthroplasty Register, Department of Orthopedic Surgery, Haukeland University Hospital
Locations (1):
- Department of Orthopeadic Surgery, Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leta TH, Gjertsen JE, Dale H, Hallan G, Lygre SHL, Fenstad AM, Dyrhovden GS, Westberg M, Wik TS, Jakobsen RB, Aamodt A, Rohrl SM, Gothesen OJ, Lindalen E, Heir S, Ludvigsen J, Bruun T, Hansen AK, Aune KEM, Warholm M, Skjetne JP, Badawy M, Hovding P, Husby OS, Karlsen OE, Furnes O. Antibiotic-Loaded Bone Cement in Prevention of Periprosthetic Joint Infections in Primary Total Knee Arthroplasty: A Register-based Multicentre Randomised Controlled Non-inferiority Trial (ALBA trial). BMJ Open. 2021 Jan 28;11(1):e041096. doi: 10.1136/bmjopen-2020-041096. PMID 33509845